CLINICAL TRIAL: NCT01132391
Title: Perianal vs Endoanal Application of Glyceryl Trinitrate 0.4% Ointment in the Treatment of Chronic Anal Fissure: Results of a Randomized Controlled Trial.
Brief Title: Perianal Versus Endoanal Application of Glyceryl Trinitrate 0.4% Ointment for Chronic Anal Fissure
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital General Universitario Elche (Other)
Responsible Party: Dr.Antonio Arroyo Sebastian, Coloproctology Unit. University Hospital of Elche
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FAC
Record Dates: First submitted 2009-09-08; First posted 2010-05-28 (Estimated); Last update posted 2010-05-28 (Estimated); Status verified 2009-09

CONDITIONS: Chronic Anal Fissure
Keywords: anal fissure; nitroglycerin; medical treatment
MeSH Terms: conditions — Fissure in Ano | interventions — Nitroglycerin; Ointments

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Endoanal application
  Interventions: Drug: Rectogesic® (glyceryl trinitrate 0.4% ointment)
- 2 (Experimental): Perianal application
  Interventions: Drug: Rectogesic® (glyceryl trinitrate 0.4% ointment)

INTERVENTIONS:
Drug: Rectogesic® (glyceryl trinitrate 0.4% ointment) — 375 mg of ointment(1,5 mg of glyceryl trinitrate ) / 12h DURING 6 MONTHS

SUMMARY:
Perianal topical nitroglycerin has been widely used as a means for avoiding surgery in patients with anal fissure. However, nitroglycerin has not been universally accepted for this application because of inconsistency of efficacy and side effects. Recent studies (Dis Colon Rectum. 2007 Apr;50(4):509-16) have demonstrated that nitroglycerin ointment products compounded by pharmacies did not meet the USP specifications for potency and/or content uniformity when filling a prescription for 0.3 percent nitroglycerin ointment. These results raise significant issues as to whether the patient is put at undue risk relative to the relief of their anal fissure pain. In addition, one study (Dis Colon Rectum. 2006 Jun;49(6):865-8) has demonstrated that intra-anal dosing of topical nitroglycerin produces a significantly greater reduction in sphincteric pressure and lower incidence of headaches than with perianal administration of the same dose of ointment.

Topical glyceryl trinitrate 0.4% ointment has been developed and tested in clinical trials and is effective in healing chronic anal fissures. It assures exactly dose and concentration of nitroglycerin.

Hypothesis: The endoanal application of exactly dose and concentration of nitroglycerin must reduced headache and the final recurrence.

The purpose of this study is:

1. Principal end-point: to compare perianal vs endoanal application of Rectogesic and evaluate the different morbidity of the two presentation

DETAILED DESCRIPTION:
inclusion criteria: chronic anal fissure. Outcome measures: recurrence and headache.

ELIGIBILITY:
Inclusion Criteria:

* Before a definitive definition of chronic anal fissure and ensuring inclusion in the study, all patients diagnosed as having chronic anal fissure based on their medical history and physical exploration were treated for a minimum of six weeks with conservative medical treatment (high residue diet, analgesics, and warm sitz baths). Chronic anal fissure was defined by the presence of a fibrous induration or exposed internal sphincter fibres.

Exclusion Criteria:

* Associated anal pathologies (incontinence, stenosis, abscess, fistula and haemorrhoids)
* Patients with associated conditions (inflammatory bowel disease, acquired immunodeficiency syndrome, tuberculosis, sexually transmitted disease and immunosuppression)
* Cardiopathy
* Headache and pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-01; Primary Completion 2009-04 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Headache (during eights weeks of treatment) | Visual analogical Score

SECONDARY OUTCOMES:
Recurrence or persistence anal fissure (six month) | Yes/No

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Arroyo, PhD, Principal Investigator
Locations (1):
- Coloproctology Unit. Elche Hospital, Elche, Alicante, Spain

REFERENCES:
- [Derived] Perez-Legaz J, Arroyo A, Moya P, Ruiz-Tovar J, Frangi A, Candela F, Oliver MI, Calpena R. Perianal versus endoanal application of glyceryl trinitrate 0.4% ointment in the treatment of chronic anal fissure: results of a randomized controlled trial. Is this the solution to the headaches? Dis Colon Rectum. 2012 Aug;55(8):893-9. doi: 10.1097/DCR.0b013e31825a9f1f. PMID 22810476 (Retraction: PMID 23652758 Madoff RD. Dis Colon Rectum. 2013 Jun;56(6):802)